CLINICAL TRIAL: NCT04561414
Title: A Prospective, Multi-center, Single-blind, Parallel, Randomized Controlled Clinical Trial (IRIS) Designed to Evaluate the Safety and Effectiveness of the LED Light Source System for Endoscope During Ureter Transillumination
Brief Title: Objective to Evaluate the Safety and Effectiveness of LED Light Source System for Endoscopy in Ureteral Radiography
Acronym: IRIS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was registered but never started.
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Stryker03
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Lower Abdominal Surgery; Pelvic Surgery
Keywords: rectal cancer; endometriosis; cervical cancer; adenomyosis; pelvic adhesion
MeSH Terms: conditions — Rectal Neoplasms; Endometriosis; Uterine Cervical Neoplasms; Adenomyosis | interventions — Endoscopes

STUDY DESIGN:
Intervention Model Description: The prospective, multi-center, single-blind, parallel, randomized controlled superiority trial design is adopted to evaluate the safety and effectiveness of the LED light source system for endoscope during ureter transillumination. The trial will be carried out in 5 centers, with the competitive grouping mode adopted. This trial will be carried out in the General Surgery Department and the Gynecology Department. Totally 120 subjects with rectal cancer, endometriosis, cervical cancer, adenomyosis and pelvic adhesion requiring operation (60 subjects for each of the test group and control group) are involved.
Who Masked: Participant
Masking Description: In this trial, single-blind method will be used, which means that the investigators know about the device used for treatment of the subjects while the subjects know nothing about it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- LED light source system for endoscope (Other): The prospective, multi-center, single-blind, parallel, randomized controlled superiority trial design is adopted to evaluate the safety and effectiveness of the LED light source system for endoscope during ureter transillumination. The trial will be carried out in 5 centers, with the competitive grouping mode adopted. This trial will be carried out in the General Surgery Department and the Gynecology Department. Totally 120 subjects with rectal cancer, endometriosis, cervical cancer, adenomyosis and pelvic adhesion requiring operation (60 subjects for each of the test group and control group) are involved. The test group use LED light source system for endoscope
  Interventions: Device: LED light source system for endoscope
- Ureteral stent (Cook Ireland Ltd.) (Other): The prospective, multi-center, single-blind, parallel, randomized controlled superiority trial design is adopted to evaluate the safety and effectiveness of the LED light source system for endoscope during ureter transillumination. The trial will be carried out in 5 centers, with the competitive grouping mode adopted. This trial will be carried out in the General Surgery Department and the Gynecology Department. Totally 120 subjects with rectal cancer, endometriosis, cervical cancer, adenomyosis and pelvic adhesion requiring operation (60 subjects for each of the test group and control group) are involved. The control group use Ureteral stent (Cook Ireland Ltd.)
  Interventions: Device: Ureteral stent (Cook Ireland Ltd.)

INTERVENTIONS:
Device: LED light source system for endoscope — The prospective, multi-center, single-blind, parallel, randomized controlled superiority trial design is adopted to evaluate the safety and effectiveness of the LED light source system for endoscope during ureter transillumination. The trial will be carried out in 5 centers, with the competitive grouping mode adopted. This trial will be carried out in the General Surgery Department and the Gynecology Department. Totally 120 subjects with rectal cancer, endometriosis, cervical cancer, adenomyosis and pelvic adhesion requiring operation (60 subjects for each of the test group and control group) are involved. The test group use LED light source system for endoscope.
  Arms: LED light source system for endoscope
Device: Ureteral stent (Cook Ireland Ltd.) — The prospective, multi-center, single-blind, parallel, randomized controlled superiority trial design is adopted to evaluate the safety and effectiveness of the LED light source system for endoscope during ureter transillumination. The trial will be carried out in 5 centers, with the competitive grouping mode adopted. This trial will be carried out in the General Surgery Department and the Gynecology Department. Totally 120 subjects with rectal cancer, endometriosis, cervical cancer, adenomyosis and pelvic adhesion requiring operation (60 subjects for each of the test group and control group) are involved. The test group use Ureteral stent (Cook Ireland Ltd.).
  Arms: Ureteral stent (Cook Ireland Ltd.)

SUMMARY:
This clinical trial is a prospective, multi-center, single-blind, parallel, randomized controlled superiority clinical trial. The trial will be carried out in 5 centers, involving 120 subjects as estimated who will be divided into the test group or control group randomly on an equal basis (each group includes 60 subjects).

This trial will be carried out in 4 stages, including the screening period, random grouping, operation date and follow-up period. In the screening period, the informed consent forms are collected and candidates are screened; after screening, the accepted subjects will be randomly divided into the control group or test group; on the operation date, the operation is carried out using the device tested; safety follow-up visit is carried out during the follow-up period.

DETAILED DESCRIPTION:
The prospective, multi-center, single-blind, parallel, randomized controlled superiority trial design is adopted to evaluate the safety and effectiveness of the LED light source system for endoscope during ureter transillumination. The trial will be carried out in 5 centers, with the competitive grouping mode adopted. This trial will be carried out in the General Surgery Department and the Gynecology Department. Totally 120 subjects with rectal cancer, endometriosis, cervical cancer, adenomyosis and pelvic adhesion requiring operation (60 subjects for each of the test group and control group) are involved. The subjects, after signing the informed consent form approved by the Ethics Committee, will be screened by the investigators. Qualified subjects who meet all the inclusion criteria and do not meet any of the exclusion criteria will be randomly divided into the control group or the test group. The subjects in the control group will accept the ureteral stent (manufacturer: Cook Ireland Ltd.) during operation. The subjects in the test group will undergo surgery using the LED light source system for endoscope and the supporting IRIS ureter kit. On the operation date, the investigators will score the performance using a scale to evaluate the resolution of the ureter in the whole process of operation. During the follow-up period, the investigators will evaluate the safety of the device based on the results of vital signs, physical examination, blood routine examination, routine urine examination, blood biochemistry, 12-lead ECG and B-mode ultrasonography of urinary system.

ELIGIBILITY:
1. Inclusion Criteria:

   1. The surgeon believes preventative placement of a ureteral stent is necessary and the target organ to be excised in the surgery is closely related to the ureter (e.g. representative specialized operations such as rectal cancer and endometriosis, cervical cancer, adenomyosis and pelvic adhesion).
   2. Age: 18 to 80 years old;
   3. All subjects voluntarily participate in the clinical trial and are asked to sign the informed consent form.
2. Exclusion Criteria:

   1. Women during pregnancy or lactation;
   2. Subjects are involved in other clinical trials at the same time; Hydronephrosis due to urinary tract obstruction; Laparotomy is expected (except for conversion to laparotomy during operation);
   3. Other conditions deemed by the investigators as unsuitable for operation;
   4. Other conditions deemed by the investigators as unsuitable for the trial (including anticipated catheterizing failure).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Resolution of the ureter in the whole operation. | in the whole process of operation
  On the operation date, the investigators will score the performance using a scale (1 very good - 10 worst outcome) to evaluate the resolution of the ureter in the whole process of operation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Principal Investigator — Beijing Friendship Hospital
Locations (4):
- China (4):
  - Beijing Chao-Yang Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Jilin University, Jilin, Changchun
  - Obstetrics&Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality